CLINICAL TRIAL: NCT03168256
Title: A Phase 3 Randomized, Double-Blind, Placebo- and Active-Controlled Study of the Efficacy and Safety of Daily CF101 Administered Orally in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: CF101 Therapy in Patients With Moderate-to-severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF101-301PS
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — CF101; N(6)-(3-iodobenzyl)-5'-N-methylcarboxamidoadenosine; apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- CF101 2mg (Experimental): CF101 2mg, orally q12 hours
  Interventions: Drug: CF101 2mg
- CF101 3mg (Experimental): CF101 3mg, orally q12 hours
  Interventions: Drug: CF101 3mg
- Apremilast 30mg (Active Comparator): Apremilast 30mg, orally q12 hours
  Interventions: Drug: Apremilast 30mg
- Placebo (Placebo Comparator): Placebo control , orally q12 hours
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: CF101 2mg — CF101 tablets, 2mg BID for 16 weeks
  Other Names: IB-MECA
  Arms: CF101 2mg
Drug: CF101 3mg — CF101 tablets, 3mg BID for 16 weeks
  Other Names: IB-MECA
  Arms: CF101 3mg
Drug: Apremilast 30mg — Apremilast tablets, 30mg BID for 16 weeks
  Other Names: Otezla
  Arms: Apremilast 30mg
Drug: Placebo Oral Tablet — Placebo tablets, BID for 16 weeks
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This trial will test the hypothesis that the administration of CF101, a novel anti-inflammatory agent, to patients with moderate to severe plaque psoriasis will relieve signs and symptoms of the disease. CF101 effect will be in comparison to apremilast in this study population

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo- and active-controlled, study in adult males and females, aged 18 to 80 years, inclusive, with a diagnosis of moderate-to-severe chronic plaque psoriasis.

Eligible subjects will be randomly assigned to CF101 2 mg, 3 mg, matching apremilast 30 mg BID, or matching placebo, in a 3:3:3:2 ratio. Blinding will be maintained using a double-dummy technique.

Medication will be taken orally BID for 32 weeks in a double-blinded fashion, with the option to continue treatment through an Extension Period to 48 weeks. Subjects initially assigned to the placebo group will be re-randomized at Week 16 to either CF101 2 mg, CF101 3 mg, or apremilast (with appropriate dose titration) in a 1:1:1 ratio and treated through Week 32, while subjects originally assigned to 1 of the active treatment groups will remain on that treatment through Week 32. The primary efficacy endpoint will be assessed at Weeks 16 and 32; at Week 32, all subjects will be offered the opportunity to remain on their assigned blinded drug through Week 48 (ie, the Extension Period of Weeks 33-48).

Disease will be assessed using PASI , static PGA , the percentage of BSA involved, and PDI. Subjects will return for assessments and a new supply of study medication at Weeks 4, 8, 12, 16, 20, 24, and 28, and for final study assessments at Week 32. For those subjects continuing into the Extension Period, efficacy and safety assessments will also occur at Weeks 36, 40, 44, and 48. PK will be assessed in a subgroup of approximately 120 subjects at Weeks 0, 8, 16, 24 and 32. PK will be assessed through sparse sampling. Assessment of whole blood A3AR expression levels will occur at Screening, Week 16, and Week 32.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 80 years of age, inclusive;
2. Diagnosis of moderate-to-severe chronic plaque-type psoriasis with BSA involvement ≥10%, as judged by the Investigator;
3. PASI score ≥12 (Appendix 3)
4. Static PGA ≥3 (Appendix 2)
5. Candidate for systemic treatment or phototherapy for psoriasis;
6. Duration of psoriasis of at least 6 months;
7. Elevated whole blood A3AR expression level, defined as ≥ 1.5-fold over a predetermined normal population standard at Screening;
8. Females of child-bearing potential must have a negative serum pregnancy test at screening;
9. Females of child-bearing potential must be willing to use 2 methods of contraception deemed adequate by the Investigator (for example, oral contraceptive pills plus a barrier method) to be eligible for, and continue participation in, the study;
10. Ability to complete the study in compliance with the protocol; and
11. Ability to understand and provide written informed consent.

Exclusion Criteria:

1. Psoriasis limited to erythrodermic, guttate, palmar, plantar, or generalized pustular psoriasis in the absence of plaque psoriasis;
2. Prior treatment with apremilast within 4 weeks prior to the Baseline visit, or contraindication to apremilast;
3. Treatment with systemic retinoids, corticosteroids, tofacitinib, or immunosuppressive agents (e.g., methotrexate, cyclosporine) within 4 weeks of the Baseline visit;
4. Treatment with a biological agent (etanercept, adalimumab, efalizumab, infliximab, ustekinumab, alefacept, secukinumab, or others, including investigational agents) within a period of time equal to 5 times its circulating half-life, or 30 days, whichever is longer, prior to the Baseline visit;
5. Treatment with high potency topical dermatological corticosteroids (Class I-III in US, Class III-IV in Europe), Vitamin D analogs, keratolytics, or coal tar (other than on the scalp, palms, groin, and/or soles) within 2 weeks of the Baseline visit;
6. Ultraviolet or Dead Sea therapy within 4 weeks of the Baseline visit, or anticipated need for either of these therapies during the study period;
7. Treatment with lithium, hydroxychloroquine or chloroquine within 2 weeks of the Baseline visit, or anticipated need for such drugs during the study period, unless dose has been stable for 3 months prior to the Screening visit and will remain stable throughout the trial;
8. Serum creatinine level greater than 1.5 times the laboratory's upper limit of normal at Screening;
9. Liver aminotransferase levels greater than 1.5 times the laboratory's upper limit of normal at Screening;
10. Electrocardiogram (ECG) at Screening shows abnormalities which, in the judgment of the Investigator, are clinically significant and could, in the judgment of the Principal Investigator, compromise subject safety;
11. Active gastrointestinal disease which could interfere with the absorption of oral medication;
12. Pregnancy, planned pregnancy, lactation, or inadequate contraception as judged by the Investigator;
13. Active drug or alcohol dependence;
14. History of depression or suicidal ideation within the past year;
15. Concomitant use of strong cytochrome P450 inducers, eg, rifampin, phenobarbital, phenytoin, carbamazepine;
16. Previous participation in a CF101 clinical trial;
17. Significant acute or chronic medical or psychiatric illness that, in the judgment of the Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study;
18. Participation in another investigational drug or vaccine trial concurrently or within 30 days prior to the Screening visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) score response of ≥75% (PASI 75) at Week 16 | 16 weeks
  Evaluate the efficacy of oral CF101 2 mg or 3 mg twice daily (BID) in patients with moderate-to-severe plaque psoriasis, compared with placebo, as determined by the proportion of subjects who achieve a Psoriasis Area and Severity Index (PASI) score response of ≥75% (PASI 75) at Week 16 (superiority)
Adverse event profile in this patient popluation | 16 weeks
  Nature, incidence and severity of treatment-emergent adverse events

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) score response of ≥50% (PASI 50) at Week 16 | 16 weeks
  Evaluate the efficacy of oral piclidenoson 2 mg or 3 mg BID, compared with placebo, as determined by the proportion of subjects who achieve PASI 50 at Week 16 (superiority);
Physician Global Assessment (PGA) | 16 weeks
  Evaluate the efficacy of oral piclidenoson 2 mg or 3 mg BID, compared with placebo, as determined by the proportion of subjects who achieve PGA score of 0 or 1 at Week 16;
Psoriasis Disability Index (PDI) | 16 weeks
  Evaluate the efficacy of oral piclidenoson 2 mg or 3 mg BID, compared with placebo, as determined by the proportion of subjects who achieve improvement on the PDI at Week 16;
CF101 PASI 75 compare to apremilast | weeks 16-32
  Evaluate the efficacy of oral piclidenoson 2 mg or 3 mg BID, compared with apremilast, as determined by the proportion of subjects who achieve PASI 75 at Weeks 16 and 32;
CF101 PGA score compare to apremilast | weeks 16-32
  Evaluate the efficacy of oral piclidenoson 2 mg or 3 mg BID, compared with apremilast, as determined by the proportion of subjects who achieve PGA score of 0 or 1, at Weeks 16 and 32;
CF101 PASI 50 compare to apremilast | weeks 16-32
  Evaluate the efficacy of oral piclidenoson 2 mg or 3 mg BID, compared with apremilast, as determined by the proportion of subjects who achieve PASI 50 at Weeks 16 and 32;
CF101 PDI improvement compare to apremilast | weeks 16-32
  Evaluate the efficacy of oral piclidenoson 2 mg or 3 mg BID, compared with apremilast, as determined by the proportion of subjects who achieve an improvement in PDI at Weeks 16 and 32;
Apremilast PASI 75 compare to placebo | weeks 16-32
  Establish assay sensitivity within this trial by comparing the efficacy of apremilast 30 mg BID with that of placebo tablets BID, as determined by the proportion of subjects who achieve PASI 75, PGA score of 0 or 1, PASI 50, and improvement in PDI at Week 16 (superiority);
Apremilast PGA compare to placebo | weeks 16-32
  Establish assay sensitivity within this trial by comparing the efficacy of apremilast 30 mg BID with that of placebo tablets BID, as determined by the proportion of subjects who achieve PGA score of 0 or 1 at Week 16;
Apremilast PASI 50 compare to placebo | weeks 16-32
  Establish assay sensitivity within this trial by comparing the efficacy of apremilast 30 mg BID with that of placebo tablets BID, as determined by the proportion of subjects who achieve PASI 50 at Week 16;
Apremilast PDI compare to placebo | 16 weeks
  Establish assay sensitivity within this trial by comparing the efficacy of apremilast 30 mg BID with that of placebo tablets BID, as determined by the proportion of subjects who achieve improvement in PDI at Week 16;
Adverse event profile of piclidenoson through the Extension Period of up to 48 weeks of treatment | 48 weeks
  Nature, incidence, and severity of treatment-emergent adverse events
Efficacy of piclidenoson, as determined by changes in PASI score, through the Extension Period of up to 48 weeks of treatment | 48 weeks
  The proportion of subjects who achieve a Psoriasis Area and Severity Index (PASI) score response of ≥75% (PASI 75) at Week 48
Determine pharmacokinetics (PK) of piclidenoson under the circumstances of this trial using sparse sampling | 48 weeks
  Serum concentration of piclidenoson
Evaluate the relationship between pre-treatment whole blood A3 adenosine receptor (A3AR) expression levels and response to piclidenoson treatment. | 16 weeks
  Explore the relationship between white blood cell (WBC) adenosine A3 receptor (A3AR) expression and treatment response, by taking WBC sample at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Michael David, MD, Principal Investigator — Rabin Medical Center
Locations (30):
- Bosnia and Herzegovina (3):
  - Clinical Centre of Republika Srpska, Banja Luka
  - University Clinical Centre Mostar, Mostar
  - Clinical Centre of Sarajevo University, Sarajevo
- Bulgaria (6):
  - "Multiprofile Hospital for Active Treatment - Pazardzhik", Pazardzhik
  - "MHAT"Rahila Angelova"AD, Department of Skin and Venereal Diseases, Pernik
  - "University Multiprofile Hospital for Active Treatment - D-r Georgi Stranski" - EAD, Pleven, Clinic of Skin and Venereal Diseases, Pleven
  - "Diagnostic-Consultative Aleksandrovska" EOOD, Sofia
  - "Diagnostic-Consultative Centre XX - Sofia" EOOD, Sofia
  - Ambulatory for Specialized Medical Help - Group Practice Dermatology - Clinic EuroDerma" OOD, Sofia
- K. Papp Clinical Research, Waterloo, Canada
- Croatia (2):
  - Clinical Hospital Center Rijeka, Rijeka
  - Sestre milosrdnice University Hospital Center, Zagreb
- Rambam Medical Center, Haifa, Israel
- Moldova (3):
  - Institutul de Cardiologie, Chisinau
  - Spitalul Clinic Municipal Nr. 3 "Sfanta Treime", Chisinau
  - Spitalul Clinic Republican, Chisinau
- Poland (6):
  - Centrum Usług Medycznych MaxMed, Bochnia
  - Gdańskim Centrum Zdrowia, Gdansk
  - All-MED Centrum Medyczne, Lodz
  - Miejski Szpital Zespolony Klinika Dermatologii Chorób Przenoszonych Drogą Płciową i Immunologii klinicznej, Olsztyn
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - ETG Zamość, ul. Szczebrzeska 11i, Zamość
- Romania (3):
  - Centrul Medical de Diagnostic si Tratament Ambulator Neomed SRL, Brasov
  - SC PELICAN Impex SRL, Oradea
  - Spitalul Clinic Județean de Urgență Sibiu, Sibiu
- Serbia (5):
  - Clinical Centre of Serbia, Belgrade
  - Clinical Centre Nis, Niš
  - Military Hospital Nis, Niš
  - General Hospital Sremska Mitrovica, Sremska Mitrovica
  - General Hospital Zajecar, Zaječar

REFERENCES:
- [Derived] Papp KA, Beyska-Rizova S, Gantcheva ML, Slavcheva Simeonova E, Brezoev P, Celic M, Groppa L, Blicharski T, Selmanagic A, Kalicka-Dudzik M, Calin CA, Trailovic N, Ramon M, Bareket-Samish A, Harpaz Z, Farbstein M, Silverman MH, Fishman P; COMFORT-1 Study Investigators. Efficacy and safety of piclidenoson in plaque psoriasis: Results from a randomized phase 3 clinical trial (COMFORT-1). J Eur Acad Dermatol Venereol. 2024 Jun;38(6):1112-1120. doi: 10.1111/jdv.19811. Epub 2024 Jan 26. PMID 38279575